CLINICAL TRIAL: NCT06813872
Title: Effectiveness of ABRYSVO® Maternal Respiratory Syncytial Virus (RSV) Vaccine Against RSV in Infants in Western Pennsylvania
Acronym: CASSATT
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3671074; CASSATT (Other: Alias Study Number)
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Viruses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Cases for the primary objective will be infants meeting the outcome definition who had any positive laboratory-confirmed RSV test from a respiratory sample collected within 10 days prior to hospital admission through 3 days after hospital admission.
  Interventions: Biological: ABRYSVO Vaccination
- Control: Controls for the primary objective will be infants meeting the outcome definition who had a laboratory-confirmed negative RSV test from a respiratory sample collected within 10 days prior to hospital admission through 3 days after hospital admission.
  Interventions: Biological: ABRYSVO Vaccination

INTERVENTIONS:
Biological: ABRYSVO Vaccination — The primary exposure of interest for the TND study is maternal history of vaccination with Pfizer's ABRYSVO vaccine during pregnancy with the infant who presented for care. Infants will be considered "exposed to ABRYSVO" if their birth parent has documented evidence of receiving ABRYSVO ≥14 days before the date of the infant's birth, during the licensed gestational age window of 32 0/7 to 36 6/7 weeks.

SUMMARY:
Globally, respiratory syncytial virus (RSV) is the leading cause of lower respiratory tract disease (LRTD) in infants and children. Pfizer has developed ABRYSVO-a bivalent RSV prefusion F protein-based vaccine (RSVpreF) composed of two prefusion F proteins to protect against both RSV-A and RSV-B. In the United States, ABRYSVO has been approved and recommended for active immunization of pregnant individuals from 320/7 to 366/7 weeks' gestational age for the prevention of LRTD and severe LRTD caused by RSV in infants from birth through 6 months of age. Post-licensure data from the United States and Argentina have also demonstrated real world effectiveness. Data from the US VISION and NVSN networks reported 79% (95% CI 55-90) and 70% (95% CI 28-88%) VE respectively against RSV-associated hospitalization among infants in the second RSV season and a study from Argentina reported 78.6% (95% CI 62.1-87.9) and 71.3% (95% CI 53.3-82.3) VE against RSV-associated LRTD leading to hospitalization among infants aged 0 to ≤3 and 0 to ≤6 months respectively.

To generate critical evidence to support vaccine policy and implementation, Pfizer will collaborate with University of Pittsburgh to study vaccine effectiveness (VE) of ABRYSVO vaccination during pregnancy against RSV-associated outcomes in infants. The study will take place in a real-world population in Western Pennsylvania over multiple seasons, beginning in the 2023-2024 season, and will use a test negative design (TND) approach.

There will be no active enrollment of study participants, no direct contact with study participants, and no collection of any primary data outside of the Standard of Care (SOC).

This study will use a TND to evaluate real-world VE of maternal ABRYSVO against RSV-associated outcomes in infants. Additionally, we will describe RSV-associated medically-attended visits for infants exposed to ABRYSVO and RSV monoclonal antibodies (e.g., Beyfortus and Enflonsia).

ELIGIBILITY:
Population included in ABYRSVO VE analyses:

1. Infants ≤ 6 months (≤ 180 days) of age on the index date.
2. Index date within the time period for data collection (approximately 01 October to 15 April in the 2023-2024, 2024-2025, 2025-2026, and 2026-2027 RSV seasons).
3. Infants born at ≥32 weeks of gestation.
4. Infants born to individuals who were expected (based on estimated date of delivery) to reach the indicated ABRYSVO vaccination window (320/7 to 366/7 weeks' gestation) during the local vaccination season.
5. Infant's EHR links to the maternal EHR.
6. Hospitalized at a UPMC facility during the RSV season (according to local hospital epidemiology) with acute respiratory tract illness symptoms meeting the protocol-defined clinical case, and for whom RSV testing results from a specimen collected 10 days prior to hospital admission through 3 days after hospital admission are known.
7. Ability to document maternal ABRYSVO receipt or not.

Population excluded from ABYRSVO VE analyses:

1. Infants who received any licensed or investigational RSV preventive product (e.g., RSV monoclonal antibodies, RSV vaccine (including investigational products or due to medication error)) since birth.
2. Born to birth parent for whom ABRYSVO vaccination status cannot be verified in the maternal EHR or Pennsylvania Immunization Electronic Registry System (PIERS) system.
3. Infants who were born to an individual vaccinated with ABRYSVO prior to the current pregnancy or vaccinated with more than one dose of ABRYSVO or vaccinated with any other licensed or investigational RSV vaccine during pregnancy.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include infants who were hospitalized with ARI, have documented RSV test results and born to an individual eligible for ABRYSVO vaccination in pregnancy based on the timing of birth relative to the local seasonal ABRYSVO vaccination program.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
RSV-positive ARI hospitalization confirmed by ³1 ARI symptom, laboratory testing, and hospitalization occurring 0 to ≤ 90 days of life during RSV season based on local epidemiology. | 0 to ≤ 90 days of life

SECONDARY OUTCOMES:
RSV-positive ARI hospitalization confirmed by ³1 ARI symptom, laboratory testing, and hospitalization occurring 0 to ≤ 180 days of life during RSV season based on local epidemiology. | 0 to ≤180 days of life
RSV-positive ARI hospitalization confirmed by ≥ 1 ARI symptom, laboratory testing, and hospitalization occurring 91 to ≤180 days of life during the RSV season based on local epidemiology | 91 to ≤180 days of life
RSV-positive ARI hospitalization with study-defined LRTD occurring 0 to ≤ 90 days of life during RSV season based on local epidemiology. | 0 to ≤90 days of life
RSV-positive hospitalization with study-defined LRTD occurring 0 to ≤180 days of life during the RSV season based on local epidemiology. | 0 to ≤180 days of life
RSV-positive ARI hospitalization with study-defined LRTD occurring 91 to ≤ 180 days of life during RSV season based on local epidemiology. | 91 to ≤ 180 days of life
Number, age and characteristics of infants whose birth parent received ABRYSVO during pregnancy who present for a medical visit (outpatient, urgent care, emergency room, hospital) and have laboratory confirmed RSV between 0 to ≤ 90 days of life | 0 to ≤90 days of life
Number, age and characteristics of infants who received Beyfortus or Enflonsia between 0 to <7 days of life who present for a medical visit and have laboratory confirmed RSV between 1 to ≤ 96 days post-B | 1 to ≤96 days post-Beyfortus/Enflonsia exposure

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671074